CLINICAL TRIAL: NCT03597321
Title: Comparative Phase II Trial of Early Prophylactic Donor Lymphocyte Infusion After Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Acute Myeloid Leukemia
Brief Title: Early Prophylactic Donor Lymphocyte Infusion After Allo-HSCT for Patients With AML
Acronym: ELIT-AML01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELIT-AML01-IPC 2017-006
Record Dates: First submitted 2018-07-16; First posted 2018-07-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Allogeneic hematopoietic stem cell transplantation; donor lymphocyte infusion
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A-DLI (Experimental): Patients will be planned to receive prophylactic Donor Lymphocyte Injection
  Interventions: Biological: prophylactic donor lymphocyte infusion (DLI)
- Arm B- No intervention (No Intervention)

INTERVENTIONS:
Biological: prophylactic donor lymphocyte infusion (DLI) — DLI will be collected from the donor by leukapheresis according to local standard procedures of each center. Cell product could be collected in one time or more, and administered fresh or after a frozen storage, according to each center's guidelines. A sufficient amount of T-cell dose should be collected to theoretically perform 3 DLI. DLI procedure will be performed according to local guidelines of each center.
  Arms: Arm A-DLI

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is a curative option for patients with acute myeloid leukemia (AML). However, transplantation related toxicity and mortality as well as the existence of HLA identical sibling donor represent major limitations. Over the 20 past years, the development of reduced intensity conditioning (RIC) regimen and the use of alternative donors allowed extending the possibility of Allo-HSCT for AML, with decreased toxicity and mortality. This invited to propose this strategy to more advanced patients, making that AML recurrence has become one of the main issues after Allo-HSCT. Thus, to develop prophylactic and preemptive strategies to minimize disease recurrence after Allo-HSCT is now the main challenge in the field. Among cellular and/or pharmacological treatments after Allo-HSCT, donor lymphocyte infusion (DLI) is probably one of the most commonly used treatments after Allo-HSCT. Indeed, DLI were reported as a potential efficient immunotherapy more than 20 years ago for the treatment of patients with leukemia relapsing after Allo-HSCT. However, most of experiences were reported in the setting of relapse after Allo-HSCT and no prospective evaluation of prophylactic DLI is available so far. Thus no strong recommendation for the use of DLI after Allo-HSCT can be made. Our study proposal would like to assess the question of prophylactic DLI efficacy, as a proof of concept of early immune intervention after Allo-HSCT. The investigators, therefore, designed a prospective multicenter randomized trial evaluating the impact of early DLI on outcome after Allo-HSCT for AML.

ELIGIBILITY:
Inclusion Criteria:

* AML in hematological complete remission at the time of inclusion
* Patient age from 18 to 70.
* Able to comply with the protocol.
* Written informed consent.
* Allogeneic stem cell transplantation from any donor except cord blood.
* Unmanipulated bone marrow or peripheral blood stem cells as graft source are allowed
* Ongoing GVHD prophylaxis using cyclosporin A at the time of inclusion.

Exclusion Criteria:

* Presence or history of grade 2 to 4 acute GVHD.
* No hematological CR of AML at the time of inclusion. CR patients positive with molecular or phenotypic minimal residual disease (MRD) can be included.
* Pregnancy/breast feeding.
* Patient considered socially or psychologically unable to comply with the treatment and the required medical follow-up.
* Concomitant uncontrolled disease and/or organ dysfunction (infection, severe heart, renal, respiratory or hepatic failure…).
* Primary or secondary graft failure.
* Previous solid organ allogeneic transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) at 2 years after randomization | 2 years
  RElpase-free survival will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test. Survival will be calculated from the date of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Raynier Devillier, MD,PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches Du Rhône, France